CLINICAL TRIAL: NCT06748560
Title: Effects of Neurodynamic Sliding Versus Eccentric Training on Lower Extremity Function, Strength and Proprioception in Athletes with Short Hamstring Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Elif Tuğçe Çil, Assistant Prof. Dr., Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOHAMMADYEDITEPESPORTTHESIS
Record Dates: First submitted 2024-12-03; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Hamstring Tightness; Hamstring Injury Prevention
Keywords: Hamstring; Tightness; Neurodynamics; Eccentric exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Eccentric training (Active Comparator): The group is consist of 13 participants who did the following treatment protocol:
  The Nordic exercise served as the foundation for the intervention, focusing on eccentric loading as participants resisted falling forward. To minimize DOMS and ensure adherence, a two-week preparatory phase of mixed concentric/eccentric leg curls using a stability ball was implemented. Following this, the gradual progression outlined by Mjolsnes et al. led to a four-week Nordic hamstring curl regimen. Weekly supervision ensured proper technique and compliance throughout the program.
  Interventions: Other: Eccentric training
- Neurodynamic sliding technique (Active Comparator): The group is consist of 14 participants who did the following treatment protocol:
  The neurodynamic sliding technique (NST) was applied to the dominant leg's sciatic nerve in the NST and ETNST groups. The technique involves alternating stress proximally and distally to promote nerve sliding. Participants performed two sets of movements-cervical flexion with knee and ankle flexion, and cervical extension with knee and ankle extension-repeated actively for 60 seconds, five times per session. Over six weeks, both groups underwent three supervised sessions per week led by an experienced researcher.
  Interventions: Other: Neurodynamics
- Eccentric training and neurodynamic sliding technique (Experimental): The group consist of 13 participants who did the following treatment protocol:
  They underwent a combined treatment incorporating both eccentric training (ET) and the neurodynamic sliding technique (NST). Participants followed the graduated Nordic hamstring exercise protocol for eccentric strengthening, alongside the nerve-sliding movements targeting the sciatic nerve. This combined approach aimed to optimize muscle flexibility, strength, and neural mobility. The interventions were performed over six weeks, with three supervised sessions per week to ensure proper execution and adherence.
  Interventions: Other: Neurodynamics; Other: Eccentric training
- Control (No Intervention)

INTERVENTIONS:
Other: Neurodynamics — Following Castellote-Caballero et al., the neurodynamic sliding technique (NST) was applied to the dominant leg's sciatic nerve in the NST and ETNST groups. The technique involves alternating stress proximally and distally to promote nerve sliding. Participants performed two sets of movements-cervical flexion with knee and ankle flexion, and cervical extension with knee and ankle extension-repeated actively for 60 seconds, five times per session. Over six weeks, both groups underwent three supervised sessions per week led by an experienced researcher.
  Arms: Eccentric training and neurodynamic sliding technique; Neurodynamic sliding technique
Other: Eccentric training — The Nordic exercise served as the foundation for the intervention, focusing on eccentric loading as participants resisted falling forward. To minimize DOMS and ensure adherence, a two-week preparatory phase of mixed concentric/eccentric leg curls using a stability ball was implemented. Following this, the gradual progression outlined by Mjolsnes et al. led to a four-week Nordic hamstring curl regimen. Weekly supervision ensured proper technique and compliance throughout the program.
  Arms: Eccentric training; Eccentric training and neurodynamic sliding technique

SUMMARY:
Hamstring strains are among the most common injuries in field sports, accounting for 10% of all team sports injuries and often leading to long-term absence from activities. Risk factors include older age, previous injuries, reduced flexibility, and strength deficits. The hamstrings play a critical role in dynamic stability and joint preservation, particularly for the hip and knee. While stretching is crucial for injury prevention, there is debate over optimal techniques.

The neurodynamic sliding technique (NST) and eccentric training (ET) are two methods that can improve flexibility and reduce injury risk. This study uniquely combines ET with NST to address hamstring tightness in athletes, aiming to evaluate their effects individually and in combination on knee muscle strength, range of motion, proprioception, and lower limb function compared to a control group.

The hypotheses examine whether these interventions differ in their impact on eccentric and concentric knee strength, the knee flexor/extensor strength ratio, range of motion, proprioception, and dynamic balance (measured via the Y Balance Test). The null hypothesis (H0) proposes no differences, while the alternative hypothesis (H1) suggests significant differences among the intervention methods.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-30 years old
2. Have a normal body mass index (BMI)
3. Have hamstring tightness as indicated by the results of an SLR examination of less than 75o (39).
4. Have hamstring tightness as indicated Active Knee Extension Test (AKET) was used to evaluate hamstring shortness. Individuals with AKET angles less than 150 degrees were considered as samples (146).
5. Ability to perform exercises.
6. Don't having plates (implants) in the lower limbs.
7. Not having a history of fracture in the lower limb (with or without realignment process).
8. Not having history of surgery to repair joint capsules, ligaments, muscles, and nerves,
9. A history of or experiencing Hernia Nucleus Pulposus (HNP).

Exclusion Criteria:

1. Receiving physical therapy or other conventional therapy in the past 6 months.
2. Absence in one of the pre- or post-test sessions.
3. Absence of more than two sessions in practice sessions.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Passive Straight Leg Raise (SLR) test | 1-2 minutes
  To measure passive hamstring flexibility, participants will lie supine on a bed with their pelvis and opposite thigh secured using straps to prevent compensatory movements. A goniometer will be positioned with its axis at the greater trochanter of the femur, the fixed arm aligned with the midaxillary line, and the moving arm along the lateral malleolus. With the knee extended and the ankle in a neutral position to avoid calf muscle stiffness, the thigh is gently flexed until hamstring tightness is felt. The straight leg's elevation angle will be measured three times, and the average will determine hamstring flexibility. Individuals with an angle less than 75° are classified as having short hamstring muscles.

SECONDARY OUTCOMES:
Knee muscle strength | 10 minutes
  Quadriceps and hamstring strength will be measured using the Biodex Pro 3 isokinetic device. Participants will sit comfortably with their trunk, pelvis, and thigh secured by straps, and the dynamometer axis aligned with the knee joint's center of rotation. After adjustments for proper positioning, the test leg will be attached to the device. Following familiarization and warm-up contractions, participants will perform maximum effort tests. Strength will be evaluated at angular speeds of 60°/s and 120°/s in both concentric and eccentric modes, with knee joint movement controlled between 0° and 90°.
Knee joint proprioception | 10 minutes
  Knee joint proprioception was assessed using the Biodex dynamometer in continuous passive motion mode at a constant speed of 5°/s. Participants sat with knees and hips bent at 90°, aligned with the dynamometer's axis, while wearing a blindfold and pneumatic boot to block visual and tactile cues. The test involved 90° of knee movement, from full extension (0°) to full flexion (90°). After practice trials, participants aimed to identify a target position (60°) during knee flexion and hit an abort button when they believed they reached it. The deviation from the target position was recorded based on three repetitions.
Y balance test | 15 minutes
  YBT test performance was assessed with a Y Balance Test Kit. Before assessment, participants were acquainted with the Y-Balance Test (YBT) by practicing on their injured limb. The YBT was performed on a platform. Throughout the task, the standing leg remained on the platform, while the other leg executed error-free maximum reach in three directions: anterior, posteromedial, and posterolateral. Maximum distances in each direction, relative to the stance leg, were measured. During the test, participants kept their hands on their waists, and each direction was repeated three times with a 10-second rest between trials.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Tuğçe ÇİL, Assistant Prof. Dr., Study Director — Physiotherapy and Rehabilitation department, Yeditepe University, istanbul, Turkey
Locations (1):
- Yeditepe university, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided